CLINICAL TRIAL: NCT06773572
Title: Efficacy of Autologous Exosomes vs Platelet-derived Growth Factors for Ovarian Regeneration in Women With Ovarian Insufficiency and Infertility: Observational, Prospective, Randomized, Comparative, Double-blind, Analytical, Prospective
Brief Title: Use of Autologous Exosomes vs Platelet Growth Factors to Regenerate the Ovary in Women With Infertility (Exosomas2024-1)
Acronym: Exosom2024-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotech Fertility C.A. (Other)
Responsible Party: Principal Investigator, Carmen Navarro, Human Reproduction Specialist, Biotech Fertility C.A.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Exosom2024-1; Eficacia en el uso de exosomas (Other: Ministerio del Poder Popular para la Salud)
Record Dates: First submitted 2024-12-22; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Female; Reproductive Techniques, Assisted
Keywords: reproductive function; exosomes; follicular function; fertility; pregnancies
MeSH Terms: conditions — Infertility, Female; Helping Behavior

STUDY DESIGN:
Intervention Model Description: An observational, prospective, randomized, comparative, double blind and analytic pilot study conducted in a fertility clinic in Caracas, Venezuela from January 2024 to September 2024, where a total of 30 patients between 38 and 46 years of age willing to become mothers underwent ovarian biostimulation procedures.
  Interventional Study Model:
  This is a quantitative correlational, inter and intra group study that aims to measure the response of the aged or resistant ovary to the contribution of platelet growth factors in activated PRP, Autologous Exosomes and their different components such as Micro-mRNA, Proteins, Sirtuins and extracellular matrix stimulants, in addition to the response to the action of the physiological solution and the trauma of ovarian puncture to reactivate the ovary, favoring the formation of new oocytes contained in the so-called Oogonia Nests.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autologous Exososomes procedure obtained from the patients' own platelets. (Active Comparator): Intraovarian injection (into the ovarian cortex) was performed over four cycles, once a month in each ovary on days 7, 8, or 9 of the menstrual cycle. Blood was drawn using the selected PRP kit; in this case, all the PRP was placed into two 20 cc syringes and filtered for exosomes using the EXOSMAT kit for autologous platelet exosomes. As a result, 5 to 6 cc of liquid composed exclusively of platelet-derived exosomes was obtained, with a concentration of 5 to 6 trillion exosomes per milliliter. Finally, 2 to 3 cc were administered to each ovary via the transvaginal route.
  Interventions: Procedure: Autologous Exososomes procedure obtained from the patients' own platelets.
- Patient group for activated platelet growth factors (Active Comparator): Intraovarian injection (into the ovarian cortex) was performed over four cycles, once a month in each ovary on days 7, 8, or 9 of the menstrual cycle. The plasma was prepared in two 5 cc syringes to administer 2 to 3 cc into each ovary (into the ovarian cortex) with the patient under sedation. The PRP was applied via the transvaginal route using a follicular aspiration needle for the PRP group.
  Interventions: Procedure: Patient group for activated platelet growth factors
- 3. Group of patients for physiological solution. (Placebo Comparator): A total of 2 to 3 cc of saline solution was administered into each ovarian cortex over four cycles, following the same protocol as the previous two groups.
  Interventions: Procedure: the control group

INTERVENTIONS:
Procedure: Autologous Exososomes procedure obtained from the patients' own platelets. — Intraovarian injection (into the ovarian cortex) was performed over four cycles, once a month in each ovary on days 7, 8, or 9 of the menstrual cycle. Blood was drawn using the selected PRP kit; in this case, all the PRP was placed into two 20 cc syringes, and the exosomes were filtered using the EXOSMAT kit for autologous platelet exosomes. A total of 5 to 6 cc of liquid composed exclusively of platelet-derived exosomes was obtained, with a concentration of 5 to 6 trillion exosomes per milliliter. Finally, 2 to 3 cc were administered to each ovary via the transvaginal route.
  Arms: Autologous Exososomes procedure obtained from the patients' own platelets.
Procedure: Patient group for activated platelet growth factors — the plasma was placed in two 5 cc injectors to place 2 to 3 cc in each ovary (in the ovarian cortex) with the patient sedated. The PRP was placed transvaginally and using a follicular aspiration needle for the PRP group. All biostimulations were performed in early follicular phase (day 7, 8 or 9) in all groups according to their assigned technique.
  Arms: Patient group for activated platelet growth factors
Procedure: the control group — Finally, the control group received 2 to 3 cc of physiological solution in each ovarian cortex for 4 cycles as the two previous groups. All these procedures were performed transvaginally under controlled surgical sedation with follicular aspiration needle in the ovarian cortex and guided by transvaginal echosonogram
  Arms: 3. Group of patients for physiological solution.

SUMMARY:
Ovarian stromal fibrosis resulting from each ovulation and due to aging is characterized by a decrease in hyaluronic acid concentrations, loss of synthesis and migration proteins CD63 and CD81, decreased miRNA125, miRNA21, miRNA132 and miRNA199. Also, enzymatic alterations affecting kinases and mitochondrial sirtuins SIRT3-5 with increased oxygen free radicals preventing the normal maintenance and development of folliculogenesis, leading to the inability to reproduce at advanced ages and accelerating the onset of pathologies secondary to the decrease of ovarian estrogens. Methodology: An observational, prospective, randomized, comparative, double-blind, analytical pilot study in 30 women between 38 and 46 years of age, with diminished ovarian reserve and who refused the egg donation procedure. Three groups were designated: one for autologous exosomes, one for PRP and one with physiological solution.

DETAILED DESCRIPTION:
METHODOLOGY AND STUDY DEVELOPMENT

This study is an observational, prospective, randomized, comparative, double-blind, and analytical investigation conducted at a fertility clinic in Caracas, Venezuela, from January 2024 to September 2024. The study involved an ovarian biostimulation or bioregeneration procedure performed on 30 patients aged 38 to 46 years with low ovarian reserve who wished to conceive using their own eggs and declined egg donation.

Patient selection criteria were based on parameters indicative of decreased ovarian reserve at the study's onset. These included hormonal levels measured on the third day of each patient's menstrual cycle: Follicle-Stimulating Hormone (FSH) greater than 12 mIU/mL, Estradiol less than 35 pg/mL, and Anti-Müllerian Hormone (AMH) less than 0.7 ng/mL. Additionally, patients had to present a total antral follicle count of fewer than five follicles across both ovaries, confirming low ovarian reserve or ovarian resistance, alongside a documented refusal to use donor eggs.

An intraovarian injection protocol was implemented based on three different treatment groups:

Autologous Exosomes obtained from the patient's platelets, Activated Platelet Growth Factors and Physiological Solution (control group).

This procedure was performed over four cycles, once per month, on days 7, 8, or 9 of menstruation. Patients were randomly assigned to one of the three groups using a randomized list managed by a trained nurse who determined allocation based on the order of arrival. The groups were distributed as follows:

Group 1: Patients receiving autologous exosomes derived from their own platelets.

Group 2: Patients receiving activated platelet growth factors. Group 3: Patients receiving a physiological solution as a placebo.

Inclusion and Exclusion Criteria

Inclusion Criteria:

* Female patients aged 38 to 46 years.
* Patients desiring to conceive.
* Patients with a Body Mass Index (BMI) between 23 and 30.
* Patients diagnosed with ovarian failure, based on the specified parameters.
* Patients refusing egg donation.
* Patients who provided informed consent after fully understanding the study.
* Patients with no active ovarian or other oncological pathologies, endometriomas, or suspected tumors.
* Patients with a platelet count exceeding 250,000 and no history of hematological diseases.
* Patients not undergoing anticoagulant therapy or presenting active infections.

Exclusion Criteria:

* Patients outside the specified age range (38-46 years).
* Patients unwilling to conceive.
* Patients with a BMI outside the 23-30 range.
* Patients without ovarian failure or who declined to participate and did not provide informed consent.
* Patients with oncological diseases or suspected tumors.
* Patients with a platelet count below 250,000.
* Patients with a history of hematological diseases, ongoing anticoagulant therapy, or active infections.

Following the initial evaluation, informed consent was obtained, and baseline laboratory tests were conducted. Blood samples were collected from each patient on the third day of their menstrual cycle before the first biostimulation to measure FSH, LH, Estradiol, AMH, and antral follicle count in each ovary. These same tests were repeated after the fourth biostimulation and before initiating fertility procedures.

All blood samples were frozen and analyzed simultaneously at a clinical laboratory in Caracas to minimize bias. Patients were advised to follow a diet free of dairy and processed carbohydrates for five days before and after each procedure. Additionally, they were encouraged to consume unflavored gelatin twice daily to enhance platelet quality.

The procedures were performed under controlled sedation in the clinic's operating room. Peripheral blood was collected from all patients using a PRP kit with separator gel, ensuring identical collection and processing protocols across all groups. Blood samples were drawn from the cubital vein using a vacutainer system under gentle compression (avoiding tourniquet use) and centrifuged at 270g for 10 minutes.

Treatment Groups:

Autologous Exosome Group: PRP was processed using the EXOSMART kit to isolate platelet exosomes. A concentrate of 6 cc containing 5-6 trillion exosomes per milliliter was obtained, and 3 cc were injected into each ovary.

Platelet Growth Factor Group: Activated PRP was prepared, and 3 cc were injected into each ovary.

Control Group: Patients received 3 cc of physiological solution injected into each ovary.

Injections were performed transvaginally using a follicular aspiration needle guided by transvaginal ultrasound. The procedures were conducted during the early follicular phase (days 7-9) under surgical sedation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 38 and 46 years of age.
* Patients with a desire to become a mother
* Patients with Body Mass Index (BMI) between 23 and 30.
* Patients with proven ovarian insufficiency, according to the parameters mentioned above.
* Patients who refuse egg donation.
* Patients with full willingness to participate in the study and who have understood and signed the informed consent.
* Patients with both ovaries without oncological pathologies, active endometriomas or suspicious ovarian or other tumors.
* Patients with platelet count over 250 thousand.
* Patients with no history of hematological diseases.
* Patients without treatment with anticoagulants.
* Patients with no active infection at the time.

Exclusion Criteria:

* Female patients outside the age range of 38 to 46 years old.
* Patients who are not willing to become mothers.
* Patients with a BMI outside the range of 23 to 30
* Patients without ovarian insufficiency
* Patients who do not wish to participate in the procedure and have not signed the informed consent form.
* Patients with suspected or diagnosed oncological diseases.
* Patients with platelet count of less than 250 thousand
* Patients with a history of hematological diseases.
* Patients with anticoagulant treatment.
* Patients with any type of active infection.

Ages: 38 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged 38 to 46 years
Enrollment: 30 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Primary Phase | Follow-up for 12 weeks for each patient.
  This study was carried out on a total of 30 patients, with an average age of 41.20 ± 2.86 years, for a minimum age of 38 and a maximum of 46 years (53.3% with ages ≤ 40 years and 46.7% aged > 40 years), with a desire to become mothers, with a previous diagnosis of resistance or ovarian failure and who also refuse egg donation.

SECONDARY OUTCOMES:
Follow-ups at birth | From the procedure to birth
  The first stage will be carried out, which is the application of the exosomes and they will be followed throughout the pregnancy until birth.

OTHER OUTCOMES:
Evaluation of the parameters of the second control that included | Monitoring during pregnancy until birth
  Count of antral follicles, collected oocytes, immature oocytes or in Metaphase I and mature oocytes or Metaphase II, fertilization rate, haploid, triploid and embryos with fragmentation greater than 35%, number of clinical pregnancies, abortions and frozen embryos

CONTACTS AND LOCATIONS:
Overall Officials: Carmen T Navarro Arrieta, Odontology, Principal Investigator — Biotech Fertility C.A.
Locations (1):
- Biotech Fertility C.A, Caracas, Venezuela

IPD SHARING:
Plan to Share IPD: Yes
We agree to share our information as long as our study is cited in each case and our copyright is respected.
Supporting Information: SAP, CSR
Time Frame: Once the study is published in the definitive journal, you will be able to obtain all the data for a period of two years after its publication.
Access Criteria: Medical specialists in Human Reproduction will be able to access the original tables and graphs of the study and inquire about the methodology and type of materials and supplies used.

REFERENCES:
- [Background] Bhatta M, Majumdar A, Ghosh U, Ghosh P, Banerji P, Aridoss S, Royal A, Biswas S, Venkatesh BT, Adhikary R, Dutta S. Sexually transmitted infections among key populations in India: A protocol for systematic review. PLoS One. 2023 Mar 13;18(3):e0279048. doi: 10.1371/journal.pone.0279048. eCollection 2023. PMID 36913427
- [Result] Melo P, Navarro C, Jones C, Coward K, Coleman L. The use of autologous platelet-rich plasma (PRP) versus no intervention in women with low ovarian reserve undergoing fertility treatment: a non-randomized interventional study. J Assist Reprod Genet. 2020 Apr;37(4):855-863. doi: 10.1007/s10815-020-01710-z. Epub 2020 Feb 7. PMID 32030554
- [Derived] Navarro C, Torrecillas Cabrera P, Teppa Garran A. Comparative analysis of the use of autologous exosomes and platelet-derived growth factors in women with premature ovarian insufficiency and infertility: A prospective, randomized, observational, analytical study. Regen Ther. 2025 Jun 30;30:309-320. doi: 10.1016/j.reth.2025.06.007. eCollection 2025 Dec. PMID 40678344